CLINICAL TRIAL: NCT01636388
Title: A Multicenter Pilot Study of Reduced Intensity Allogeneic Stem Cell Transplantation Followed by Adoptive Cellular Immunotherapy With Donor Derived Latent Membrane Protein (LMP) Specific-CTLs in Patients With Epstein-Barr Virus (EBV)Positive Refractory or Recurrent Hodgkin Lymphoma
Brief Title: Allogeneic Stem Cell Transplantation With Adoptive Immunotherapy in Epstein-Barr Virus Positive Recurrent/Refractory Hodgkins Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding ended
Sponsor: New York Medical College (Other)
Collaborators: Children's National Research Institute (Other); Baylor College of Medicine (Other); M.D. Anderson Cancer Center (Other); City of Hope Medical Center (Other); Johns Hopkins University (Other); Ohio State University (Other); University of Utah (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-553
Record Dates: First submitted 2012-06-26; First posted 2012-07-10 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Hodgkins Lymphoma
Keywords: Relapsed Hodgkins Lymphoma; Refractory Hodgkins Lymphoma; Allogeneic Stem Cell Transplantation; Adoptive Immunotherapy; Cellular Therapy; Cytotoxic T cell lymphocytes
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Stem Cell Transplantation (Experimental): Reduced intensity conditioning and allogeneic stem cell transplant from EBV positive HLA matched sibling or unrelated adult donor combined with post AlloSCT allogeneic donor derived LMP specific cytotoxic T-lymphocyte (CTL) infusions in EBV positive patients with poor risk Hodgkin Lymphoma.
  Interventions: Biological: allogeneic donor derived LMP specific cytotoxic T-lymphocyte

INTERVENTIONS:
Biological: allogeneic donor derived LMP specific cytotoxic T-lymphocyte — LMP CTLs will be give at 3 timepoints post allogeneic stem cell transplantation around days 60 to 100, then 30 days apart for the next 2 infusions.

SUMMARY:
The investigators intend to utilize reduced intensity conditioning and allogeneic stem cell transplant from EBV positive HLA matched sibling or unrelated adult donor combined with post AlloSCT allogeneic donor derived LMP specific cytotoxic T-lymphocyte (CTL) infusions in EBV positive patients with poor risk Hodgkin Lymphoma. One of three reduced intensity conditioning regimens predetermined at each institutional center of the Childhood, Adolescent and Young Adult Lymphoma Cell Therapy Consortium (LCTC) will be utilized for related or matched unrelated adult donor allogeneic transplant followed by donor LMP specific CTL infusion for three doses post AlloSCT. The investigators hypothesize that the addition of donor derived LMP specific CTLs will be safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

Patient must be 45 years of age or less.

Patient or the patient's legally authorized guardian must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects), and must sign an informed consent in accordance with the institutional policies approved by the U.S. Department of Health and Human Services.

Patients should have been off other investigational therapy for one month prior to entry in this study.

Patient must have adequate organ function as below

Adequate renal function defined as:

Serum creatinine <2.0 x normal, or Creatinine clearance or radioisotope GFR > 40 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range

Adequate liver function defined as:

Total bilirubin <2.0 x normal; and SGOT (AST) or SGPT (ALT) <5.0 x normal

Adequate cardiac function defined as:

Shortening fraction of >27% by echocardiogram

Hodgkin Lymphoma with either of the following:

Primary induction failure (failure to achieve initial CR) and/or primary refractory disease.First relapse ; Early relapse (within 12 months off therapy) (excluding those who received no therapy or radiation therapy only for initial therapy); Late relapse (greater than 12 months off therapy). Only patients with recurrent Stage III or IV disease and/or those with B symptoms at relapse (all other late relapses are excluded); Second relapse; Third relapse.

History of prior ablative auto HSCT or ineligible for an ablative auto HSCT or ≥25% residual disease after at least two reinduction chemotherapy cycles.

EBV seropositive IgG HLA matched family or unrelated donor (MUD) HLA matched family donor (6/6 or 5/6) or matched unrelated adult donor (MUD) (7/8 or 8/8) All patients entered into the study ideally will have tumor tissue from the original diagnostic specimen and/or relapse reviewed centrally for confirmation of Hodgkin lymphoma. If no specimen is available, local pathology report documenting EBV positivity is acceptable. Appropriate immunophenotyping to confirm the diagnosis will be performed. In addition, in situ hybridization for EBV (LMP1, and/or EBER positivity) will be performed. All central morphologic analysis and immunohistochemical/insitu hybridization staining will be performed in the laboratory of Sherrie Perkins and Rodney Miles at the University of Utah.

Exclusion Criteria:

Patients with HD with 4th or greater CR, PR, and/or SD are ineligible. Patients with rapidly progressive disease (PD) unresponsive to reinduction chemo, radio, or immunotherapy are ineligible.

EBV negative Hodgkin Lymphoma. Patients who don't have an eligible donor (outlined in 7.0) are ineligible. Women who are pregnant are ineligible. Negative pregnancy test in women of childbearing age is required.

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  The number of serious adverse events associated with administering allogeneic HLA matched donor derived LMP specific-CTLs in CAYA with EBV-associated refractory/relapsed HL following reduced intensity conditioning (RIC) and allogeneic HSCT will be monitored to determine the safety of this treatment.
Toxicity | 1 year
  The number of adverse events associated with administering allogeneic HLA matched donor derived LMP specific-CTLs in CAYA with EBV-associated refractory/relapsed HL following reduced intensity conditioning (RIC) and allogeneic HSCT will be monitored to determine the toxicity of this treatment.

SECONDARY OUTCOMES:
Feasibility | 1 year
  Good Manufacturing Practice (GMP) production and shipping of HLA matched donor derived LMP specific-CTLs to multiple sites in various geographic regions of the US following RIC and allogeneic HSCT will be monitored to assess the feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States